CLINICAL TRIAL: NCT04345887
Title: The Effect of Spironolactone on Oxygenation in Covid-19 ARDS Patients
Brief Title: Spironolactone in Covid-19 Induced ARDS
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Olcay Dilken, Dr., Istanbul University - Cerrahpasa
Other Study IDs: 10042020
Record Dates: First submitted 2020-04-10; First posted 2020-04-15 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Respiratory Distress Syndrome, Adult
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Canrenoic Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Spironolactone: 2 x 100 mg spironolactone
  Interventions: Drug: Spironolactone 100mg
- Placebo: 2 x 1 placebo
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Spironolactone 100mg — 2x100 mg spironolactone for 5 consecutive days
  Groups: Spironolactone
Drug: Placebo oral tablet — 2 x1 placebo tablet
  Groups: Placebo

SUMMARY:
This study intended to evaluate the effects of commonly used diuretic, spironolactone, on oxygenation in covid-19 ARDS patients.

ELIGIBILITY:
Inclusion Criteria:

* Hemodynamically stable
* Hypoxemia, i.e. p/f <150
* Admitted to ICU within 48 hours
* Not moribund has a life expectancy greater than 24 hours

Exclusion Criteria:

* Age criteria
* Pregnancy
* Unwillingness to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients admitted to the ICU due to Covid-19 ARDS requiring diuretic
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-05-05 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-07-05 (Actual)

PRIMARY OUTCOMES:
p/f ratio | 5 days
  improvement in oxygenation

SECONDARY OUTCOMES:
SOFA | 5 days
  improvement in SOFA Score

CONTACTS AND LOCATIONS:
Overall Officials: Yalim Dikmen, Study Director — Prof
Locations (1):
- Istanbul University-Cerrahpaşa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vaduganathan M, Vardeny O, Michel T, McMurray JJV, Pfeffer MA, Solomon SD. Renin-Angiotensin-Aldosterone System Inhibitors in Patients with Covid-19. N Engl J Med. 2020 Apr 23;382(17):1653-1659. doi: 10.1056/NEJMsr2005760. Epub 2020 Mar 30. No abstract available. PMID 32227760